CLINICAL TRIAL: NCT03852875
Title: The Impact of Patient Knowledge on Treadmill Performance
Brief Title: Impact of Pt Knowledge on TM Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REB112887
Record Dates: First submitted 2018-12-13; First posted 2019-02-25 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Cardiac Rehabilitation; Stress Testing
Keywords: Cardiac Rehabilitation; Stress Testing; Education
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Experimental): Patients in the experimental arm will receive a 1-on-1 education session to review the their CR participation. As part of the discussion about their CR participation, these patients will also receive feedback on their intake exercise stress test.
  Interventions: Other: Education
- Control (Sham Comparator): Patients in the Control arm will receive a 1-on-1 education session to review the their CR participation. As part of the discussion about their CR participation, these patients will NOT receive feedback on their intake exercise stress test.
  Interventions: Other: Control

INTERVENTIONS:
Other: Education — Same
  Arms: Education
Other: Control — Same
  Arms: Control

SUMMARY:
The primary outcome of the Cardiac Rehabilitation (CR) program at St Joseph's Hospital is change in performance on an exercise stress test. Patients complete an exercise stress test when they enter and exit the CR program. An improvement in stress test performance reflects an improvement in physical fitness, but is also associated with better long-term health outcomes (e.g. reducing the chance of having to go back to hospital; lower likelihood of dying). While physical fitness has the strongest impact on stress test performance, other factors can also affect the test result. We expect that informing patients about their baseline stress test result will improve their exit treadmill performance. This intervention may be a simple and cost-effective method of increasing motivation among patients to do their best on the exit test

DETAILED DESCRIPTION:
Cardiac rehabilitation (CR) is a class 1 or "strong" recommendation in contemporary clinical practice guidelines following percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG) after a myocardial infarction (MI)[1-6]. The CR program at St. Joseph's Hospital is a 6 month intensive program focusing on education, exercise and lifestyle changes [7, 8] with the goal of helping the patient improve their functional capacity. The Canadian Cardiovascular Society has set a benchmark of a 0.5 MET increase in functional capacity as one of 5 Quality Indicators (QIs) of CR programs [7, 8]. Quality indicators seek to quantify the quality of CR in a well-defined and evidence based manner. To measure the improvement in functional capacity, CR participants complete an exercise stress test at intake to and exit from the CR program. The improvement on this test is one of the main outcomes of a CR program while illustrating the impact of the CR program on the individual.

Performance on the exercise stress test can be used to predict coronary heart disease and all-cause mortality risk levels in patients [9]. Patients with higher aerobic fitness have a favourable cardiovascular risk factor profile [9]. Obtaining an accurate measure of the patient's fitness levels during the exit stress test is essential to creating an appropriate future care plan. In order to optimize results on the exit stress test, the other contributing factors to performance must be optimized as well.

Past studies suggest that patients may exercise at a lower metabolic intensity without feedback [10]. This result shows the potential increase in performance on the exercise stress test if patients are given feedback. Given that participant feedback, knowledge of results and motivation can all have an effect on performance, we are interested to see if providing additional information to our patients about their performance on their previous (intake) stress test will have an impact on their performance at the exit test.

When the patient learns about their previous performance, they will be better informed of their capacity and should be inclined to improve results at their exit test. If the other contributing factors surrounding one's performance on the treadmill are optimized, the cardiac care team will have a better understanding of the patient's true fitness. This will help the team propose an accurate plan for the future direction of the patient's care

ELIGIBILITY:
Inclusion Criteria:

* Patients who completing the St Joseph's Hospital CR Program
* Patients exiting the CR program with available results (ECG and metabolic) from their intake assessment
* Patients who are able to comprehend the educational intervention at their exit from CR
* Willing to participate in research and sign informed consent

Exclusion Criteria:

* Patients who decline participation
* CR patients without available results from intake assessment
* Patients who, based on the clinical judgement of the attending physician, have some transitory health issue (e.g. cold, infection, biomechanical issues) that may impact their performance on the TM test.
* Patients who are unable to perform the treadmill test

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Change in METs | Intake assessment is at T=0 (baseline). Exit assessment is at approximately 6 months (exit)
  Improvement in Treadmill Performance as expressed in TM-derived METs
Change in VO2peak | Intake assessment is at T=0 (baseline). Exit assessment is at approximately 6 months (exit)
  Improvement in Treadmill Performance as measured by metabolic testing (VO2 measurement) during Treadmill test

CONTACTS AND LOCATIONS:
Overall Officials: Neville Suskin, MbCHb, Principal Investigator — St Joseph's Hospital
Locations (1):
- St Joseph's Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No